CLINICAL TRIAL: NCT00956826
Title: Continuous Fetal Monitoring During Vacuum Delivery an Addition of a New Device
Brief Title: Continuous Fetal Monitoring During Vacuum Delivery
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Hadassah Medical Organization (Other)
Responsible Party: David Mankuta, Hadassah University Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: fetal monitoring vaccum; FMV123
Record Dates: First submitted 2009-07-19; First posted 2009-08-11 (Estimated); Last update posted 2009-08-11 (Estimated); Status verified 2009-08

CONDITIONS: Vacuum Delivery
Keywords: electrode vacuum delivery

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Electrode added to device (Experimental): With an electrode and a regular vacuum device
  Interventions: Device: Agit Vacuum

INTERVENTIONS:
Device: Agit Vacuum — With an electrode and a regular vacuum device
  Other Names: Agit Vaccum

SUMMARY:
The investigators have added an additional electrode to the vacuum device for birth in which they can monitor the fetus during delivery.

DETAILED DESCRIPTION:
The investigators have added an additional electrode to the vacuum device for birth in which they can monitor the fetus during delivery. The electrode is a standard one inserted in the vacuum device.

ELIGIBILITY:
Inclusion Criteria:

* All fetuses at vacuum delivery

Exclusion Criteria:

* None

Ages: 1 Day to 1 Day | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2009-09; Primary Completion 2010-04 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
Quality of fetal heart rate monitoring in both arms | 12 month

CONTACTS AND LOCATIONS:
Overall Officials: David Mankuta, MD, Study Chair — Hadassah
Locations (1):
- Hadassah Ein Kerem, Jerusalem, Israel